CLINICAL TRIAL: NCT06498856
Title: Saline Infusion Test in Hyponatremia
Acronym: SITH
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Hormone Laboratory, Aker University Hospital, Oslo, Norway (Other)
Responsible Party: Principal Investigator, Jacob Winther, MD, PhD, Head of Endocrinology department, University Hospital, Akershus
Other Study IDs: 23/12081
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Hyponatremia
Keywords: Arginine vasopressin; Copeptin; Antidiuretic hormone; Saline infusion test; Fluid- and volume regulation; Renin; Aldosterone
MeSH Terms: conditions — Hyponatremia; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with hypoosmolar hyponatremia: Patients admitted to hospital with hypo-osmolar hyponatremia with uncertain primary cause. Eligible patients will receive a standardized intravenous infusion of isotonic saline.
  Interventions: Other: Isotonic saline infusion

INTERVENTIONS:
Other: Isotonic saline infusion — Volume expansion with one liter of isotonic saline intravenously over two hours.

SUMMARY:
Observational study of biochemical volume biomarker levels in response to a standardized intravenous isotonic saline infusion in patients with hyponatremia.

DETAILED DESCRIPTION:
Hyponatremia (low plasma sodium concentration) is a common electrolyte disorder among hospitalized patients that can lead to complications such as gait instability, falls and mental changes. Both hyponatremia itself and overly rapid correction of hyponatremia may lead to brain damage.

There are several underlying causes of hyponatremia that require different treatment strategies. Specifically, hypovolemia is treated with fluid infusion while other common causes such as the syndrome of inappropriate diuresis (SIAD) and hypervolemic conditions need fluid restriction. In clinical practice, it can be challenging to identify the main cause of hyponatremia due to overlapping diagnosis and unreliable diagnostic tools, typically leading to a timely trial and error approach to therapy.

A saline infusion test (SIT) is often used to diagnose hypovolemic hyponatremia. To our knowledge, the test has never been validated, but relies on the rationale that the sodium concentration will increase more with saline infusion in hypovolemia than in other causes of hyponatremia. Typically, one liter of isotonic saline is infused intravenously and an arbitrarily set cut-off for sodium increase is used to indicate hypovolemia. As the response of sodium depends on several factors that affects the renal free water excretion capacity, this measure may not be the most accurate nor the most efficient. Another, more direct, approach could be to measure the change in biochemical markers of circulating volume in response to the volume expansion that comes with saline infusion. We will measure several different biomarkers before, during and after a standardized isotonic saline infusion in patients hospitalized with hyponatremia. Based on the results, we hope to develop a more precise tool for the differential diagnosis of hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Plasma sodium 120-130 mmol/L
* Effective osmolality (2 x plasma sodium + plasma glucose) < 275 milliosmol/L
* Age > 18 years

Exclusion Criteria:

* Intensive care unit (ICU) admission
* Adequate sodium correction rate: > 4 mmol/L last 24 hours
* Primary polydipsia: urine osmolality < 100 mOsm/L
* Hypertonic saline therapy
* Adrenal insufficiency
* Severe heart failure: ejection fraction < 35 % or clinical suspicion of decompensated heart failure
* Ascites grade 3 (marked abdominal distention and discomfort)
* Chronic renal failure stage 4 or 5: estimated glomerular filtration rate < 30
* Failure to submit informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with hyponatremia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Copeptin plasma levels | 240 minutes
  Changes in copeptin levels in response to isotonic saline infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jacob A Winther, MD,PHD, Study Director — University Hospital, Akershus

IPD SHARING:
Plan to Share IPD: Undecided